CLINICAL TRIAL: NCT00063830
Title: ISIS 2302-CS27, Phase 2, Double-Blinded, Controlled Study of Four Dosing Regimens of Alicaforsen (ISIS 2302) Enema, an Antisense Inhibitor of ICAM-1, for the Treatment of Patients With Mild to Moderate Active Ulcerative Colitis
Brief Title: ISIS 2302-CS27, A 6-Week, Placebo-Controlled Clinical Study to Evaluate the Effectiveness of Alicaforsen (ISIS 2302) in Patients With Mild to Moderate Active Ulcerative Colitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Purpose: Treatment
Other Study IDs: ISIS 2302-CS27
Record Dates: First submitted 2003-07-07; First posted 2003-07-08 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2007-10

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — alicaforsen

INTERVENTIONS:
Drug: Alicaforsen

SUMMARY:
This is a multi-center trial in the US and Europe to test the safety, efficacy and tolerability of alicaforsen (ISIS 2302), a new type of drug called an antisense drug, in patients with mild to moderate active Ulcerative Colitis (UC). Alicaforsen is designed to reduce the production of a specific protein, called ICAM-1, a substance that plays a significant role in the increase of inflammation and is likely to be involved in inflammatory bowel diseases such as ulcerative colitis. The ISIS 2302-CS27 study will compare four dosing regimens and determine the minimum effective dose of alicaforsen enema in UC patients over six weeks as compared to a placebo enema. (The probability of receiving active formulation is 4:1). The primary objective of this study is to evaluate the percentage reduction in DAI at Week 6.

ELIGIBILITY:
Inclusion Criteria

Patients must meet the following criteria at screening to be eligible for enrollment:

* Age greater than or equal to 18 years
* Diagnosis of left-sided ulcerative colitis of at least 6 months duration
* Current left-sided flare, defined as activity in the colon 5-50 cm from the anal verge, extending at least 15 cm proximal to the anal verge and confirmed by endoscopic evaluation within 14 days of baseline visit.
* Baseline DAI score of 4-10 including abnormal endoscopic score
* On at least one or more of the following treatments for ulcerative colitis prior to baseline visit:

  1. Stable background oral mesalamine therapy for greater than or equal to 30 days, and/or
  2. Stable background mercaptopurine for greater than or equal to 60 days prior to baseline, and/or
  3. Stable azathiprine therapy for greater than or equal to 60 days prior to baseline
* Written informed consent prior to performing screening evaluations.

Exclusion Criteria

Patients who meet any of the following criteria at screening are not eligible for enrollment:

* Bowel stricture, toxic megacolon, colonic dysplasia, adenoma or carcinoma
* Patients with pancolitis
* Uncontrolled hematologic, renal, hepatic, metabolic, psychiatric, CNS, pulmonary or cardiovascular disease, or sufficient level of disease that could interfere with the patient's ability to comply with protocol participation
* Enteric pathogens or presence of Clostridium difficile toxin in stool
* History of colon resection
* Major surgical procedure within one month of baseline visit
* Steroid or mesalamine enema within 14 days of baseline visit
* Systemic steroids (including ACTH) within 30 days of baseline visit
* Tumor necrosis factor-alpha (TNF-α) inhibitor treatment within 90 days of baseline visit
* Non-steroidal anti-inflammatory agents (NSAIDs), including cyclooxygenase-2 (COX-2) inhibitors, within 14 days of baseline visit
* Methotrexate, cyclosporin or thalidomide within 90 days of baseline visit
* Any active infection currently requiring treatment
* Malignancy within 5 years except for squamous cell or basal cell cancers of the skin
* Current infectious, ischemic, or immunological disease with gastrointestinal involvement
* ISIS 2302 treatment within 12 months of baseline visit
* Treatment with an investigational or off-label drug within 90 days of screening or currently in long-term follow up for another investigational treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04-03 (Actual); Primary Completion 2004-10-11 (Actual); Study Completion 2004-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sacramento, California, United States